CLINICAL TRIAL: NCT04639999
Title: Impact of MIgalastat TheRApy on CaRdiac Function in patiEnts With Fabry's Cardiomyopathy (MIRACRE-Fabry Trial)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-1038
Record Dates: First submitted 2020-11-10; First posted 2020-11-23 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10cc blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fabry's disease: Fabry's disease patients who were confirmed by enzyme assay and gene study
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — LV vortex flow in Echocardiography

SUMMARY:
This is an observational study. No treatment or intervention will be assigned to the subjects. All patients will receive full standard of care concomitant medication for the treatment of their cardiac condition. 20 patients with genetically confirmed Anderson-Fabry disease who have a plan to start Migalastat will undergo 2D strain, diastolic stress echocardiography, LV vortex flow analysis, and CMR at baseline and after 2 year of treatment with Migalastat for follow-up.

DETAILED DESCRIPTION:
1. Objectives - to evaluate the impact of chaperone therapy on LV diastolic function and flow in patients with Fabry's cardiomyopathy using LV 2D strain, diastolic stress echocardiography, LV vortex flow and CMR.
2. Primary/Secondary Endpoint

   A. Primary endpoint:

   - Change of peak exercise E/E' by diastolic stress echocardiography, global longitudinal strain and LV vortex flow parameters at 2 year follow up.

   B. Secondary endpoints:
   * Changes of extracellular volume by CMR (T1 mapping) at 2 year follow up
   * Evaluation of the degree of the resting LV diastolic function
   * Evaluation of global and regional LV strain
   * Other echo-parameters; LV mass index at baseline, 2 year follow up, reduction of peak exercise E/E prime at 2 year follow up
   * Changes of quality of life using questionnaire
   * Change of peak VO2, exercise time, AT by diastolic stress echocardiography at 2 year follow up
   * Change in T1 baseline (myo, ms) & T1 baseline (blood, ms) T1 postcontrast (myo, ms) & T1 baseline (blood, ms) by CMR
3. Study Methods -Study Design: This is an observational study. No treatment or intervention will be assigned to the subjects. All patients will receive full standard of care concomitant medication for the treatment of their cardiac condition. 20 patients with genetically confirmed Anderson-Fabry disease who have a plan to start Migalastat will undergo 2D strain, diastolic stress echocardiography, LV vortex flow analysis, and CMR at baseline and after 2 year of treatment with Migalastat for follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 16 ~ 70 years with Fabry's disease who were confirmed by enzyme assay and gene study
2. Patients who have LV hypertrophy in 2D echocardiography (end diastolic septum and posterior wall thickness ≥12mm) or Patients who present with cardiac changes (indicative of disease progression such as decreased global longitudinal strain on 2D strain echocardiography or low native T1 mapping on cardiac MRI) even without LV wall thickness of ≥12mm
3. Patients provided with the written, informed consent to participate in this study

Exclusion Criteria:

1. Contraindication for chaperone therapy (Migalastat)
2. Patients who cannot perform supine bicycle stress echocardiography, contrast echocardiography or cardiac MRI
3. Hemodynamically significant valvular heart disease or arrythmias
4. History of acute myocardial infarction or congestive heart failure with reduced LV ejection fraction of less than 35%
5. CVA in the prior 6 months
6. Scheduled or planned surgery in the next 6 months
7. Chronic liver cirrhosis
8. Allergy to contrast agent (Definity®, Lantheus Medical Imaging, North Billerica, MA, USA)

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 16 ~ 70 years with Fabry disease confirmed by enzyme assay and gene test
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change of peak exercise E/E' by diastolic stress echocardiography | 2 years
Change of global longitudinal strain | 2 years
Change of LV vortex flow parameters | 2 years

SECONDARY OUTCOMES:
Changes of extracellular volume by CMR (T1 mapping) | 2 years
Evaluation of the degree of the resting LV diastolic function | 2 years
Evaluation of global and regional LV strain | 2 years
Evaluation of LV mass index | 2 years
Evaluation of reduction of peak exercise E/E prime | 2 years
Changes of quality of life using Short Form 36 | 2 years
Change of peak VO2 by diastolic stress echocardiography | 2 years
Change of exercise time by diastolic stress echocardiography | 2 years
Change of AT by diastolic stress echocardiography | 2 years
Change in T1 baseline (myo, ms) & T1 baseline (blood, ms) T1 postcontrast (myo, ms) & T1 baseline (blood, ms) by CMR | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Geu-Ru Hong, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided